CLINICAL TRIAL: NCT03274830
Title: A Post Market Clinical Follow-up Study With the aneXys Cup
Status: Active, not recruiting | Type: Observational
Sponsor: Mathys Ltd Bettlach (Industry)
Responsible Party: Sponsor
Other Study IDs: 1602_V03_10042019
Record Dates: First submitted 2017-08-24; First posted 2017-09-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: primary osteoarthritis; secondary osteoarthritis; femoral head fracture; necrosis
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aneXys: cases with aneXys cup and Mathys hip stem
  Interventions: Device: aneXys

INTERVENTIONS:
Device: aneXys — 150 patients with the aneXys cup

SUMMARY:
The purpose of the study is the evaluation of the clinical and radiological short- to long-term safety and performance of the aneXys cup. The data will be used for an ongoing evaluation of the product safety and performance.

DETAILED DESCRIPTION:
Prospective observational multicenter case series providing short-term migration results and long-term post-market clinical data on the safety and performance of the aneXys cup. The study includes patients undergoing primary total hip arthroplasty. In total 100 patients in 3 clinics will be included. In each clinic 10-57 consecutive patients shall be included. In addition, to meet the regulatory requirements, a total of minimum 20 cases with screw fixation shall be included in the study.

Clinical and radiological follow-up (FU) is planned after 6-12 weeks, 6 months, 1, 2, 5, 7 and 10 years. An additional FU at 3 years is planned to apply for an ODEP (Orthopaedic Data Evaluation Panel) rating.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (signed by participant and investigator)
* Primary implantation
* Suffer from primary or secondary osteoarthritis of the hip, femoral head and neck fractures or necrosis of the femoral head. In all cases a stable anchoring of the implant has to be possible.
* Age at inclusion: between 18 and 75 years old
* Willing to participate in the follow-up examinations
* Complete recovery is expected

Exclusion Criteria:

* Missing informed consent form (signed by participant and investigator)
* Known or suspected non-compliance (e.g. drug or alcohol abuse)
* Enrolment of the investigator, his/her family, employees and other dependent persons
* Patients younger 18 years old
* Revision surgery
* Presence of sepsis or malignant tumours
* ASA (American Society of Anesthesiologists) Classification >3
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Cup migration after 2 years | 2 years
  The primary endpoint will be the radiographic evaluation of the acetabular cup migration based on performed EBRA measurements 2 years after surgery.

SECONDARY OUTCOMES:
Harris Hip Score | 10 years
  The secondary endpoint will be the determination of the clinical outcome using the Harris Hip Score.
Visual analogue scale vor pain | 10 years
  The secondary endpoint will be the determination of the clinical outcome using the Visual analogue scale for pain.
Visual analogue scale for satisfaction | 10 years
  The secondary endpoint will be the determination of the clinical outcome using the Visual analogue scale for satisfaction.
The Western Ontario and McMaster Universities Osteoarthritis Index | 10 years
  The secondary endpoint will be the determination of the clinical outcome using the WOMAC.

OTHER OUTCOMES:
Osteolysis | 6-12 weeks - 10 years
  The first endpoint of interest is the occurrence of osteolysis around the cup.
Lucent lines | 6-12 weeks - 10 years
  The second endpoint of interest is the occurrence of lucent lines around the cup.
Complications | post-op - 10 years
  The first safety endpoint will be the number of complications with respect to the investigational product.
Revisions | post-op - 10 years
  The second safety endpoint will be the number revisions with respect to the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Roth, Prof., Principal Investigator — Universitätsklinik Leipzig
Locations (3):
- Germany (3):
  - DRK Kliniken Berlin | Köpernick, Berlin
  - DRK Kliniken Berlin | Westend, Berlin
  - Universitätsklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No